CLINICAL TRIAL: NCT04994093
Title: Creating an Innovative AI-based (Artificial Intelligence) IN SILICO TECHNOLOGY TCRact to Launch a NEW SERVICE for Designing and Optimizing T-cell Receptors (TCR) for Use in Cancer Immunotherapies
Brief Title: Creating an Innovative AI-based Technology TCRact for Designing and Optimizing T-cell Receptors (TCR) for Use in Cancer Immunotherapies
Status: Completed | Type: Observational
Sponsor: Ardigen (Industry)
Collaborators: National Center for Research and Development, Poland (Other)
Responsible Party: Sponsor
Other Study IDs: TCRact; POIR.01.01.01-00-0019/20 (Other Grant/Funding Number: The National Centre for Research and Development)
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Colon Cancer; Cancer
Keywords: Immunology; TCR; FFPE; PBMC; Colon Cancer; Immuno-Oncology; Cancer; Oncology
MeSH Terms: conditions — Colonic Neoplasms; Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — stool, biopsy (FFPE) and peripheral blood samples (PBMC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COLON CANCER: This cohort will consist of 100 patients with Colon Cancer.
  Interventions: Other: Collection of blood (PBMC), biopsy (FFPE) and stool samples.

INTERVENTIONS:
Other: Collection of blood (PBMC), biopsy (FFPE) and stool samples. — Patients receiving routine treatment financed by the Polish National Health Fund (NFZ).

SUMMARY:
The PROJECT OBJECTIVE is to create an innovative AI-based (Artificial Intelligence) IN SILICO TECHNOLOGY for the design and optimization of T-cell receptors (TCRs) capable of recognizing specific tumor antigens presented on Human Leukocyte Antigen (HLA). The technology will be based on bioinformatics (including molecular modelling) and artificial intelligence (including predictive, generative and optimization models). PROJECT TASKS are dedicated to the implementation of individual technological components (including the database necessary for their preparation) and to performing IN VITRO evaluation rounds to optimize the technology.

Integration, within an IN SILICO TECHNOLOGY, of processes which currently require huge amounts of in vitro laboratory experiments that are necessary for bringing new TCR-based cancer immunotherapies into clinical trials:

* finding appropriate TCRs targeting cancer neoantigen presented on a HLA molecule (pHLA)
* testing for potential TCR toxicity (targeting self antigens presented on healthy tissues)
* optimization of pHLA:TCR binding affinity and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of advanced resectable colorectal cancer (Active stage II, III or IV)
* Histopathologically confirmed as adenocarcinoma
* Age 18 or over
* Being able to understand and sign the Informed Consent Form (ICF)
* Qualification for resection within 3 months from W0 or condition after primary tumor resection, not longer than 5 years from surgery

Exclusion Criteria:

* Mucinous colorectal adenocarcinoma
* Canal and anal edge cancer,
* Adenocarcinoma of the appendix,
* Patients treated with neoadjuvant therapy or radiation therapy in the 3 months prior to study enrollment.
* Patients treated with systemic chemotherapy in the 3 months prior to study enrollment.
* Histopathological diagnosis other than adenocarcinoma
* Remission
* History of inflammatory bowel diseases
* Pregnancy
* HIV infection
* Active infection with hepatitis B and C viruses
* Leukocytopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving routine treatment.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
Finding appropriate TCRs targeting cancer neoantigen presented on a HLA molecule (pHLA) | Inclusion
Testing for potential TCR toxicity (targeting self antigens presented on healthy tissues) | Inclusion
Optimization of pHLA:TCR binding affinity and toxicity | Inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Sklodowska-Curie National Research Institute of Oncology, Krakow, Poland

REFERENCES:
- [Derived] Bujak J, Klek S, Balawejder M, Kociniak A, Wilkus K, Szatanek R, Orzeszko Z, Welanyk J, Torbicz G, Jeckowski M, Kucharczyk T, Wohadlo L, Borys M, Stadnik H, Wysocki M, Kayser M, Slomka ME, Kosmowska A, Horbacka K, Gach T, Markowska B, Kowalczyk T, Karon J, Karczewski M, Szura M, Sanecka-Duin A, Blum A. Creating an Innovative Artificial Intelligence-Based Technology (TCRact) for Designing and Optimizing T Cell Receptors for Use in Cancer Immunotherapies: Protocol for an Observational Trial. JMIR Res Protoc. 2023 Jul 13;12:e45872. doi: 10.2196/45872. PMID 37440307